CLINICAL TRIAL: NCT01506102
Title: Determination of Thromboelastography Values in Pregnancy and After Delivery
Brief Title: Thromboelastography During and After Delivery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Città di Roma Hospital (Other)
Responsible Party: Principal Investigator, Silvia Stirparo, Staff Anesthesiologist, Città di Roma Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: TEM-A in pregnancy
Record Dates: First submitted 2012-01-05; First posted 2012-01-09 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2012-01

CONDITIONS: Delivery Uterine
MeSH Terms: interventions — Thrombelastography

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Thromboelastography — Thromboelastography during labor and after delivery
  Other Names: TEM-A automated thromboelastometer

SUMMARY:
The purpose of this study is to establish reference values for thromboelastography (TEM-A) in healthy pregnant women during labor and 2 hours and 24 hours after delivery.

DETAILED DESCRIPTION:
Previous, preliminary investigations by using thromboelastography, confirmed that pregnancy is a hypercoaguable state which remains in the first 24 hours postdelivery. Unfortunately results obtained by the existing studies that attempted to establish reference values for TEG suffer considerable bias.

The aim of this study will be to determine the range values for thomboelastography in pregnant women. Since there is no available information on the expected distribution of the outcome, a sequential design will be used. The main endpoint of the analysis will be a reliable estimate for the outcome expected in healthy women after labor. The investigators will state their target estimate as being reliable when the ratio between the estimate and its standard error is smaller than 2.

During labor, 2 hours after delivery and 24 hours postpartum, a venous blood sample will be taken from eligible women for thromboelastographic determination. Whole blood nonadditive TEM will be performed on the TEM-A automated thromboelastometer (Framar Biomedica,Rome, Italy) to obtain the four classical TEM parameters: reaction (R) time, k time, alpha angle and maximum amplitude (MA).

Inclusion criteria Healthy parturients in labor Exclusion criteria parturients who will eventually had: operative or instrumental vaginal delivery, estimated blood loss greater than 500 mL, the occurrence of II and III degree perineal lacerations, any coagulation disorder or anticoagulant therapy

ELIGIBILITY:
Inclusion Criteria:

* healthy parturients in labor

Exclusion Criteria:

* parturients with coagulation defects or anticoagulant therapy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2011-11; Primary Completion 2012-05 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
TEM-A automated thromboelastometer, Framar Biomedica,Rome, Italy | 24 hours postpartum
  To determine the physiological reference individual values of maternal thromboelastography TEM-A during labor, immediately afeter delivery and in the postpartum period.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Stirparo, MD, Principal Investigator — Città di Roma Hospital
Locations (1):
- Città di Roma Hospital, Roma, Roma, Italy